CLINICAL TRIAL: NCT02736851
Title: Home-Based Telemedicine Management of Patients Affected by Chronic Neck Pain
Brief Title: Telemedicine to Manage Chronic Neck Pain at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Bernardo Gialanella, Coordinator, Fondazione Salvatore Maugeri
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Delibera 6863,CTS 7 April 2009
Record Dates: First submitted 2016-03-16; First posted 2016-04-13 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Adherence
Keywords: disability; home; stretching exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Usual care
- Home-based telemedicine group (Active Comparator): Nurse-tutor support at home for 6 months
  Interventions: Other: Home-based telemedicine group

INTERVENTIONS:
Other: Home-based telemedicine group — All patients referring to the rehabilitation service as out-patients underwent in-hospital a specific exercise program for the neck. Patients are instructed individually by a physical therapist to perform several types of exercises and, from the first rehabilitation session, are encouraged to exercise regularly at home. Written and illustrated material reporting home exercises is provided to all patients.
  At the end of out-rehabilitation program, according to a randomization list, patients are randomized in 2 groups and those included in a Home-Based Telemedicine (HBT) program are followed up by a nurse tutor at home for a 6-month period.
  Arms: Home-based telemedicine group

SUMMARY:
The aim of the study is to investigate if a home-based structured physician-directed, nurse-managed telemedicine program can increase adherence to a home exercise program and decrease neck pain and disability.

The study is carried out in 100 consecutive patients with chronic non-specific neck pain.

All patients referred to a rehabilitation Institute for an out-.patient visit complete a stretching exercise program and are instructed and encouraged to perform exercises regularly once at home. At the end of the rehabilitation, the patients are randomized into two groups of 50 patients each. Patients of the first Group are allocated to a home-based telemedicine (HBT), while those of the second group receive only the recommendation to continue exercising at home (Control group). The HBT intervention consists of fortnightly scheduled phone calls to patients over the 6-month course of the study. A nurse-tutor encourages the patient to perform regularly physical activity and prescribes exercises.

Adherence to home exercises is evaluated 15 days and 6 months after the end of the outpatient rehabilitation, while pain intensity and neck disability are assessed and compared in the two groups at entry and 6 months after the end of the outpatient rehabilitation .

DETAILED DESCRIPTION:
Systematic reviews have concluded that exercises taught individually and prescribed to be performed at home, are effective in decreasing neck pain and avoiding recurrence of neck pain (re-exacerbations) if patients adhere to the home exercise program. Conversely, inadequate adherence to a home-based exercise program reduces the treatment's efficacy. Telemedicine is already employed in many fields of medicine to evaluate health status, treatment, education, and to monitor patients' care needs but not in management of the patients with chronic neck pain. Studies available in the literature have not yet clearly defined if a phone surveillance program is effective in decreasing pain in these patients. Conversely, we think that telemedicine may be a useful tool for physicians in management of chronic neck pain because it can increase adherence to home exercises program thus reducing neck pain and disability in these patients. To verify this hypothesis we perform this prospective randomized controlled study.

The study is performed in 100 consecutive patients with chronic non-specific neck pain referred to the outpatient facility of our Rehabilitation Department.

Patients have to be > 18 years and with neck pain duration more than 6 months. Exclusion criteria are: pain duration < 6 months, cognitive deficit, history of fracture or operations around the neck region, presence of inflammatory rheumatic diseases, neurological diseases that could lead to neck pain, infections or tumors, pregnancy, previous rehabilitation for neck pain undergone within the last 12 months, and inability to attend all exercise sessions of our outpatient rehabilitation program.

All patients have to complete, as outpatients, an exercise program consisting of 10 sessions, spread over a 2-week period (5 days/week), and including six stretching exercises for the neck.

Patients are instructed individually by a physical therapist on how to perform each exercise and, after the first rehabilitation session, are encouraged to exercise regularly at home. Written and illustrated material explaining the home exercises are provided to all patients.

At the end of the outpatient rehabilitation program, patients are randomized (using a randomization list provided by the statistical consultant) into two groups of 50 patients each. Patients of the first group are allocated to a home-based telemedicine (HBT) program for 6 months (HBT group), while those of the second group receive only recommendations to continue the exercises at home (Control group).

The HBT intervention consists of fortnightly scheduled phone calls to patients over the 6-month course of the study. A nurse-tutor collects information on: disease status, pain, disability, prodromal symptoms of exacerbation, number of home exercise sessions performed, and use of non-steroidal anti-inflammatory drugs. In consultation with the physiatrist, the nurse gives advice on solutions for persistent pain and any symptoms of exacerbation. The patient is always encouraged to perform regularly the physical activity and the exercises prescribed. The physiatrist is involved as a second-opinion consultant.

The patients are evaluated at entry and 6 months after the end of the outpatient rehabilitation by the same qualified physiatrist. At entry, scales of demonstrated reliability, validity and sensitivity are administered to assess comorbidity (evaluated with Cumulative Illness Rating Scale-Geriatrics), pain severity (10-point analogue scale), neck range of motion (manual goniometer), and neck disability (Neck Disability Index). Adherence to home exercises is evaluated 15 days and 6 months after the end of the outpatient rehabilitation and is self-reported.

Differences in adherence to home exercises, pain intensity and neck disability, between baseline and 6-month follow up, are assessed and compared in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* chronic non-specific neck pain duration more than 6 months.

Exclusion Criteria:

* pain duration less than 6 months
* willingness to sign the informed consent form (unable to read or write)
* cognitive deficit (e.g. Alzheimer disease or senile dementia)
* patient unable to attend all sessions of exercises
* inflammatory rheumatic diseases
* history of fracture or operations around the neck region
* neurological diseases that may lead to neck pain, infections or tumours
* pregnancy
* rehabilitation sessions for neck pain since less than 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in Adherence as assessed by number of exercise sessions/week | Change between 15 days and 6 months after the end of the outpatient rehabilitation
  Number of exercise sessions/week

SECONDARY OUTCOMES:
Change in Pain | Change between entry and 6 months after the end of the outpatient rehabilitation
  Evaluation by a Visual Analogue Scale (VAS)
Change in Disability | Change between entry and 6 months after the end of the outpatient rehabilitation
  Evaluation by the Neck Disability Index

CONTACTS AND LOCATIONS:
Overall Officials: Simonetta Scalvini, MD, Study Director — Fondazione Salvatore Maugeri

IPD SHARING:
Plan to Share IPD: Yes
The research was supported by a grant from Lombardy Region. A final report was provided to Lombardy Region.

REFERENCES:
- [Result] Gialanella B, Ettori T, Faustini S, Baratti D, Bernocchi P, Comini L, Scalvini S. Home-Based Telemedicine in Patients with Chronic Neck Pain. Am J Phys Med Rehabil. 2017 May;96(5):327-332. doi: 10.1097/PHM.0000000000000610. PMID 27584139